CLINICAL TRIAL: NCT00997542
Title: A Double-blind, Placebo-controlled, Cross-over Study of the Effects of Allopurinol on Oxidative Metabolism, Peripheral Blood Flow and Immune Function in Patients With Advanced Chronic Heart Failure (CHF).
Brief Title: Allopurinol in Chronic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart and Lung Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 97-044
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Heart Failure; Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol
  Arms: Allopurinol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to discover whether the inhibition of the xanthine oxidase with allopurinol leads to a reduction of the production of oxygen free radicals in patients with CHF and thereby improves characteristics of oxydative metabolism, peripheral blood flow, immune function and functional status.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male and at least 21 years of age.
* The patient has clinical evidence of heart failure: a) reduced ejection fraction (≤40%) or cardiomegaly on CXR or left ventricular impairment on echocardiography (LVEDD ≥60mm), b) stable clinical condition and medication for at least 1 month prior to the study.
* No history of unstable angina, myocardial infarction or stroke within 3 months prior to the study.
* The patient is receiving full conventional medical therapy for heart failure (ACE inhibitor or angiotensin II blocker, diuretics etc.).
* The patient is willing and capable of complying with the requirements of this protocol.
* The patient has provided written informed consent .

Exclusion Criteria:

* The patient has any life-threatening disease, other than heart failure (including patients with known, or suspected, myocarditis or with automatic implantable cardioverter/defibrillators).
* The patient has an active malignancy of any type, or history of a malignancy (Patients who have a history of basal cell carcinoma that has been surgically removed are acceptable). Patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years prior to study enrolment are also acceptable.
* The patient has had a heart transplant.
* The patient has severe renal disease (S-Creatinine >300 μmol/l), severe liver disease (ASAT or ALAT > 3 times of upper limit of normal range), rheumatoid arthritis, or complains of gout.
* The patients has received allopurinol therapy previously or if he is known to suffer from gout (acutely or chronically).
* The patient has an exercise capacity of > 20 ml/kg/min (treadmill, Bruce protocol) or is in functional NYHA class I.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)

PRIMARY OUTCOMES:
postischemic peak peripheral blood flow

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Fravel MA, Ernst ME. Management of gout in the older adult. Am J Geriatr Pharmacother. 2011 Oct;9(5):271-85. doi: 10.1016/j.amjopharm.2011.07.004. Epub 2011 Aug 17. PMID 21849262